CLINICAL TRIAL: NCT07263984
Title: SEPTUM-D Project: Diagnosis in Patients With a Uterine Septum
Brief Title: Added Value of Three-dimensional Transvaginal Ultrasound (3D TVUS) and Gel Infusion Sonography (3D GIS) Compared With Magnetic Resonance Imaging (MRI) in the Diagnosis of Patients With Suspicion of a Uterine Septum.
Acronym: SEPTUM-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2025-0219; T002825N (Other Grant/Funding Number: FWO)
Record Dates: First submitted 2025-11-14; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Uterine Septum
Keywords: Uterine septum; Diagnosis; Three-dimensional transvaginal ultrasound; Magnetic Resonance Imaging; Gel Infusion Sonography
MeSH Terms: conditions — Septate Uterus; Disease | interventions — Magnetic Resonance Imaging; Surveys and Questionnaires

STUDY DESIGN:
Masking Description: Central readers of US and MRI images
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspicion of a uterine septum on two-dimensional transvaginal ultrasound (Experimental): Patients with suspicion of a uterine septum on two-dimensional transvaginal ultrasound
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Three-dimensional transvaginal ultrasound; Diagnostic Test: Three-dimensional transvaginal Gel Infusion Sonography; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — MRI of the pelvis
Diagnostic Test: Three-dimensional transvaginal ultrasound — Three-dimensional transvaginal ultrasound
Diagnostic Test: Three-dimensional transvaginal Gel Infusion Sonography — Three-dimensional transvaginal Gel Infusion Sonography
Other: Questionnaires — Questionnaires

SUMMARY:
The goal of this clinical trial is to investigate the added value of three-dimensional transvaginal ultrasound (3D TVUS) and gel infusion sonography (3D GIS) for diagnosing a partition in the uterus (uterine septum) in comparison to magnetic resonance imaging (MRI). The main question it aims to answer is:

How well do 3D TVUS and 3D GIS detect a uterine septum compared to MRI?

Participants will receive 3D TVUS/ 3D GIS and MRI, and will complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 45 years
* With suspicion of a uterine septum on routine 2D TVUS
* Who are willing to give informed consent

Exclusion Criteria:

* Women aged below 18 years and over 45 years
* Prior definitive diagnosis of a uterine septum or other congenital uterine anomaly
* Prior surgery in relation to a uterine septum
* Cervical (unilateral) aplasia
* Vaginal aplasia
* Untreated obstructive vaginal septum
* Any co-morbidity that is found to interfere with the uterine measurements required in the study
* Contraindications for MRI
* Not willing or not possible to undergo transvaginal ultrasound
* Pregnancy at the time of inclusion
* Wish to conceive between inclusion and last diagnostic intervention
* Visual or pathological evidence of cervical, uterine or ovarian malignancy
* Patients with an intrauterine device (by mistake), who are not willing to remove this device before the start of the diagnostic interventions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of three-dimensional transvaginal ultrasound (3D TVUS) for the diagnosis of a uterine septum compared with MRI | Within 12 weeks after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium